CLINICAL TRIAL: NCT01617629
Title: An Open-Label Safety Trial of Cvac (Autologous Dendritic Cells Pulsed With Recombinant Human Fusion Protein Coupled to Oxidized Polymannose) for Epithelial Ovarian Cancer Patients Who Have Progressed During the CAN-003 Study
Brief Title: Ovarian Cancer Vaccine for Patients Who Have Progressed During the CAN-003 Study
Acronym: CAN-003X
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prima BioMed Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAN-003X
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-11

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Cvac
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — CCV-AV protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cvac Treatment Group (Experimental): Participants received Epithelial Mucin Surface Antigen 1 (MUC1) Dendritic Cell Vaccine (Cvac) treatment.
  Interventions: Biological: MUC1 Dendritic Cell Vaccine (Cvac)

INTERVENTIONS:
Biological: MUC1 Dendritic Cell Vaccine (Cvac) — The recommended dosing regimen for CAN-003X was every 4 weeks for the first 3 doses and then every 12 weeks for 3 doses, for a total of 6 doses over 44 weeks (Regimen A, applicable to CAN-003 observational Standard of Care patients and CAN-003 Cvac patients that have progressed prior to the fourth dose of Cvac).
  Participants who received more than 3 doses of Cvac in CAN-003 continued with the CAN-003 dosing schedule (Regimen B; Cvac every 4 weeks for a total of 7 doses and then every 8 weeks for 3 doses, for a total of 10 doses over approximately 48 weeks).

SUMMARY:
The purpose of this trial is to assess the safety profile of Cvac for epithelial ovarian cancer patients who were enrolled in the Cvac clinical trial CAN-003 and are no longer eligible for study participation due to disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥ 18 years old with histologically confirmed Stage III or IV epithelial ovarian, primary peritoneal, or fallopian tube cancer who were enrolled in CAN-003
* Able and willing to undergo mononuclear cell (MNC) collection (if required for patients who do not have available Cvac doses)
* Were enrolled in CAN-003 and met protocol criteria for progressive disease
* Wish to remain in the study and, in the investigator's judgment, the potential benefit of Cvac treatment outweighs the risk
* Must be non-pregnant and, if of childbearing potential, must use adequate birth control (hormonal or barrier method of birth control or abstinence) for the duration of the study and for 3 months after study completion
* Able to provide written informed consent
* White blood cell count (WBC) ≥ 3.0 K/μL, absolute neutrophil count ≥ 1.5 K/μL, hemoglobin ≥ 9.0 g/dL, and platelets ≥100,000/mm^3

Exclusion Criteria:

* Pregnant or breastfeeding
* Other medical conditions which preclude study participation, in the opinion of the investigator
* Receiving treatment with any other investigational product

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidy Gray, MD, Principal Investigator — University of Washington; James Mason, MD, Principal Investigator — Scripps Cancer Center; Peter Eisenberg, MD, Principal Investigator — Marin Cancer Care; Giuseppe Del Priore, MD, Principal Investigator — Indiana University School of Medicine; Fernando Recio, MD, Principal Investigator — Collaborative Research Group; Jeffery Goh, MBBS, FRACP, Principal Investigator — Greenslopes Private Hospital
Locations (6):
- United States (5):
  - Marin Cancer Care, Inc., Greenbrae, California
  - Scripps Cancer Center, La Jolla, California
  - Collaborative Research Group, Boca Raton, Florida
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - University of Washington Medical Center, Seattle, Washington
- Greenslopes Private Hospital, Greenslopes, Queensland, Australia

REFERENCES:
- [Background] Apostolopoulos V, McKenzie IF. Cellular mucins: targets for immunotherapy. Crit Rev Immunol. 1994;14(3-4):293-309. doi: 10.1615/critrevimmunol.v14.i3-4.40. PMID 7538768
- [Background] Apostolopoulos V, McKenzie IF, Pietersz GA. Breast cancer immunotherapy: current status and future prospects. Immunol Cell Biol. 1996 Oct;74(5):457-64. doi: 10.1038/icb.1996.76. PMID 8912009
- [Background] Desai J, Mitchell P, Loveland B, et al. A phase I trial of dendritic cells pulsed with MUC1 peptide in patients with solid tumours. Proc ASCO 2002; 21:15b (A1868).
- [Background] Apostolopoulos V, Karanikas V, Haurum JS, McKenzie IF. Induction of HLA-A2-restricted CTLs to the mucin 1 human breast cancer antigen. J Immunol. 1997 Dec 1;159(11):5211-8. PMID 9548459
- [Background] Grossi M, Quinn MA, Thursfield VJ, Francis PA, Rome RM, Planner RS, Giles GG. Ovarian cancer: patterns of care in Victoria during 1993-1995. Med J Aust. 2002 Jul 1;177(1):11-6. doi: 10.5694/j.1326-5377.2002.tb04616.x. PMID 12088472
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Background] Liu PY, Alberts DS, Monk BJ, Brady M, Moon J, Markman M. An early signal of CA-125 progression for ovarian cancer patients receiving maintenance treatment after complete clinical response to primary therapy. J Clin Oncol. 2007 Aug 20;25(24):3615-20. doi: 10.1200/JCO.2006.09.4540. PMID 17704410
- [Background] Meyer T, Rustin GJ. Role of tumour markers in monitoring epithelial ovarian cancer. Br J Cancer. 2000 May;82(9):1535-8. doi: 10.1054/bjoc.2000.1174. PMID 10789720
- [Background] Ozols RF, Rubin SC, Thomas G, et al. Epithelial ovarian cancer. In: Hoskins WJ, Perez CA, Young RC, eds. Principles and Practice of Gynecologic Oncology, 4th ed. Philadelphia: Lippincott Williams & Wilkins. 2005:919-922.
- [Background] Rustin GJ, Nelstrop AE, Bentzen SM, Bond SJ, McClean P. Selection of active drugs for ovarian cancer based on CA-125 and standard response rates in phase II trials. J Clin Oncol. 2000 Apr;18(8):1733-9. doi: 10.1200/JCO.2000.18.8.1733. PMID 10764434
- See also: Related Info from Sponsor's Web Site — http://primabiomed.com.au/investor/presentations.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with ovarian cancer who participated in CAN-003 [NCT01068509] and had disease progression were enrolled in CAN-003x in Australia and the United States from December 2011 to April 2014.
Groups:
- Cvac Treatment Group: Participants received Epithelial Mucin Surface Antigen 1 (MUC1) Dendritic Cell Vaccine (Cvac) treatment.
  MUC1 Dendritic Cell Vaccine (Cvac): The recommended dosing regimen for CAN-003X was every 4 weeks for the first 3 doses and then every 12 weeks for 3 doses, for a total of 6 doses over 44 weeks (Regimen A, applicable to CAN-003 observational Standard of Care patients and CAN-003 Cvac patients that have progressed prior to the fourth dose of Cvac).
  Participants who received more than 3 doses of Cvac in CAN-003 continued with the CAN-003 dosing schedule (Regimen B; Cvac every 4 weeks for a total of 7 doses and then every 8 weeks for 3 doses, for a total of 10 doses over approximately 48 weeks).
Period: Overall Study
Arm/Group | Cvac Treatment Group
Started | 9
Completed | 3
Not Completed | 6
Not completed — Death | 2
Not completed — Investigator's Clinical Judgement | 1
Not completed — Reason Not Specified | 1
Not completed — Participant Withdrew Consent | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who enrolled in the study.
Groups:
- Cvac Treatment Group: Participants received MUC1 Dendritic Cell Vaccine (Cvac) treatment.
  MUC1 Dendritic Cell Vaccine (Cvac): The recommended dosing regimen for CAN-003X was every 4 weeks for the first 3 doses and then every 12 weeks for 3 doses, for a total of 6 doses over 44 weeks (Regimen A, applicable to CAN-003 observational Standard of Care patients and CAN-003 Cvac patients that have progressed prior to the fourth dose of Cvac).
  Participants who received more than 3 doses of Cvac in CAN-003 continued with the CAN-003 dosing schedule (Regimen B; Cvac every 4 weeks for a total of 7 doses and then every 8 weeks for 3 doses, for a total of 10 doses over approximately 48 weeks).
Arm/Group | Cvac Treatment Group
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a study drug, whether or not considered related to the drug. A SAE is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect or is a medically important event.
Time Frame: First dose of study vaccine to 30 days past last dose (Approximately 1 Year)
Population: Safety Population included all participants who enrolled in the study.
Measure: Number; unit: participants
Arm/Group | Cvac Treatment Group
Number analyzed (Participants) | 9
participants
  Adverse Events | 7
  Serious Adverse Events | 2

2. Other Pre Specified Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization until death from any cause.
Time Frame: 2 years
Population: Due to the few patients, Overall Survival could not be calculated.
Arm/Group | Cvac Treatment Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: First dose of study vaccination to 30 days past last dose (Approximately 1 Year)
Arm/Group | Cvac Treatment Group
All-Cause Mortality (participants affected / at risk) | 2/9
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cvac Treatment Group (N=9)
Incarcerated hernia (General disorders) | 1
Wound complication (Injury, poisoning and procedural complications) | 1
Disease progression (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cvac Treatment Group (N=9)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Lymph node pain (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Blepharospasm (Eye disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Influenza like illness (General disorders) | 1
Injection site pruritus (General disorders) | 1
Oedema peripheral (General disorders) | 1
Ear infection (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Gastric infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Abnormal dreams (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For study centers in Australia, no publication of the study results may be made until publication of the results of the study from all centers or until 2 years after study completion, whichever is sooner. For study centers in the USA, no submission for publication or public disclosure of the results by will be made until the results from all centers have been received and analyzed by the sponsor, or the multi-center study has been terminated or abandoned at all centers.